CLINICAL TRIAL: NCT06314386
Title: SAIA-TB: Using the Systems Analysis and Improvement Approach (SAIA) to Prevent TB in Rural South Africa
Brief Title: Systems Analysis and Improvement Approach to Prevent TB
Acronym: SAIA-TB
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Boston University (Other); University of Washington (Other); Medical Research Council, South Africa (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 23.139.01; R01NR020866 (NIH)
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Tuberculosis; TPT; TB - Tuberculosis
Keywords: tuberculosis
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Crossover Cluster
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exposed (Other): Clinics are considered exposed after intensive SAIA-TB intervention, implementation phase, and maintenance phase.
  Interventions: Other: Systems Analysis and Improvement Approach for TB (SAIA-TB)
- Unexposed (No Intervention): Clinics are considered unexposed prior to the initiation of SAIA-TB in their clinic

INTERVENTIONS:
Other: Systems Analysis and Improvement Approach for TB (SAIA-TB) — The Systems Analysis and Improvement Approach for TB (SAIA-TB) is a five-step systems analysis and iterative improvement cycle intervention which will be implemented by clinic staff with support from study personnel in intervention clinics. Components of the intervention include TB cascade analysis, patient flow mapping and continuous quality improvement, aimed to incrementally optimize TB screening, evaluation, diagnosis, TB preventive therapy and TB disease treatment initiation, successful treatment, and TB-free survival among the population at the intervention clinics.
  Arms: Exposed

SUMMARY:
This randomized trial uses the evidence-based Systems Analysis and Improvement Approach (SAIA) adapted for tuberculosis (SAIA-TB) to assess the comprehensive tuberculosis (TB) care cascade across 16 clinics in rural Eastern Cape, South Africa to improve patient outcomes. The aims of this study are to:

* Evaluate the effectiveness of SAIA-TB use in clinics on TB cascade outcomes for TB patients and with high-risk contacts
* Determine the drivers of SAIA-TB implementation success or failure across clinics

The investigators hypothesize that SAIA-TB implementation will lead to a 20% increase in each of: TB screening, TB preventive treatment initiation, and TB disease treatment initiation during the 18-month intervention period.

DETAILED DESCRIPTION:
This four-wave stepped wedge crossover cluster randomized trial will assess the effectiveness of the SAIA-TB intervention (Aim 1). A total of 16 clinics in four municipalities within the Sarah Baartman-district, Eastern Cape, South Africa will be included. The SAIA-TB intervention will be implemented at the clinic level. Public sector clinic staff and clinic managers, supported by study personnel, will deliver the intervention over an 18-month implementation phase, followed by a 12-month maintenance phase led by clinic managers without additional study personnel support, to provide evidence on intervention impact under ideal circumstances, as well as sustained effect over time. Aim 2 will consist of interviews and using the organization readiness for implementing change (ORIC) with facilities early in SAIA-TB implementation (within 3 months of initiating the intervention) to identify clinic-level attributes that affect intervention adoption. Additionally, the Consolidated Framework for Implementation Research (CFIR) will guide data collection and interpretation related to implementation, assess ﬁdelity to intervention protocol, describe intervention adaptations when integrated into routine management systems, and identify clinic-level determinants of successful SAIA-TB implementation. Recurrent measurement of structural readiness and implementation dose (as a function of quality and quantity) at the clinic level will inform guidance on essential structural needs to implement SAIA-TB. The trial will culminate in a dissemination package, summarizing results and providing implementation guidance to support scale-up.

ELIGIBILITY:
Aim 1:

1. Inclusion Criteria for clinics:

   * Location in the municipalities of Dr. Beyers Naude, Blue Crane Route, Makana, Ndlambe, Sundays River Valley, Kou-Kamma, or Kouga within the Sarah Baartman district, Eastern Cape, South Africa
   * Within 2 hours' drive to Gqeberha, where the study office is located
   * Only one clinic per town/area/location to ensure a mix of rural, semi-rural, semi urban
   * Clinic capacity/Patient volume > 700 total outpatient attendees per month (8,400 patients per year)
   * Staff size of at least 5 employees with a mixture of at least 2 professional nurses, 1 or 2 pharmacist/pharmacy technicians, at least 1 data capturer, a social worker, and multiple community health workers who are clinic-based or part of ward-based outreach teams.
   * Must have an acting Clinic Manager
2. Exclusion Criteria for clinics:

   * Clinic managers and/or staff are unwilling to participate

Aim 2:

1. Inclusion Criteria:

   * 18 years and older
   * Frontline clinical and/or managerial staff, district-level TB management
   * Ability to provide informed consent
2. Exclusion Criteria:

   * Under age 18
   * Unwilling to provide informed consent

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19560 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
TB Screening | 18 months
  The proportion of individuals screened with WHO TB symptom screen in the target population
Linkage to care for TB disease treatment | 18 months
  The proportion of individuals initiating TB disease treatment among those with a positive diagnostic evaluation
Linkage to care for TB preventive treatment | 18 months
  The proportion of individuals initiating TB preventive treatment among those with a negative diagnostic evaluation and eligible for TPT

SECONDARY OUTCOMES:
Successful TB Prevention Treatment (TPT) Outcome | 18 months
  The proportion of individuals who complete TB Prevention Treatment (TPT) among those who initiate TPT
Successful TB Outcome | 18 months
  The proportion of individuals cured or completing treatment for TB disease among those who initiate TB treatment
TB Evaluation | 18 months
  The proportion of individuals receiving a diagnostic evaluation among those with a positive screening
TB Diagnosis | 18 months
  The proportion of individuals diagnosed with TB among those who completed a diagnostic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Brittney J van de Water, PhD, Principal Investigator — Boston College
Locations (16):
- South Africa (16):
  - Addo Clinic, Addo
  - Lukhanyiso Clinic, Addo
  - Kwa-Nonqubela Clinic, Alexandria
  - Marselle Clinic, Boesmansriviermond
  - Masakhane Clinic, Hankey
  - Humansdorp Clinic, Humansdorp
  - Pellsrus Clinic, Jeffrey's Bay
  - Joubertina CHC, Joubertina
  - Louterwater Clinic, Joubertina
  - Twee Riviere Clinic, Joubertina
  - Kareedouw Clinic, Kareedouw
  - Kenton On Sea Clinic, Kenton on Sea
  - Kirkwood Clinic, Kirkwood
  - Moses Mabida Clinic, Kirkwood
  - Imizamo Yetho Clinic, Patensie
  - Nkwenkwezi Clinic, Port Alfred

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van de Water BJ, Brooks MB, Matji R, Ncanywa B, Dikgale F, Abuelezam NN, Mzileni B, Nokwe M, Moko S, Mvusi L, Loveday M, Gimbel S. Systems analysis and improvement approach to optimize tuberculosis (SAIA-TB) screening, treatment, and prevention in South Africa: a stepped-wedge cluster randomized trial. Implement Sci Commun. 2024 Apr 16;5(1):40. doi: 10.1186/s43058-024-00582-z. PMID 38627799